CLINICAL TRIAL: NCT06031103
Title: Clinical Efficacy of Mini-Percutaneous Nephrolithotomy Versus Retrograde Intrarenal Surgery for the Management of Upper Urinary Tract Calculus (1-2.5 cm) in Children ≤10 Years of Age
Brief Title: Clinical Efficacy of Mini-PCNLversus RIRS for the Management of Upper Urinary Tract Calculus (1-2.5 cm)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pediatric renal stones
Record Dates: First submitted 2023-08-19; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-08

CONDITIONS: Stone, Kidney
Keywords: Pediatric stones; retrograde intrarenal surgery; mini-per-cutaneous nephrostomy
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- childhood urolithiasis treated with mini PCNL Procedure (Active Comparator): pediatric patients with upper urinary tract calculus treated with mini-PCNL procedure
  Interventions: Procedure: mini-PCNL procedure
- childhood urolithiasis treated with RIRS Procedure (Active Comparator): pediatric patients with upper urinary tract calculus treated with mini-PCNL procedure
  Interventions: Procedure: RIRS procedure

INTERVENTIONS:
Procedure: mini-PCNL procedure — Mini-PCNL
  . A 12 Fr rigid nephroscope and a Holmium:YAG laser as energy source was used for surgery Percutaneous renal puncture was achieved with an 18 Ga needle after displaying renal collecting system with contrast material. and tract dilatation was achieved using Amplatz dilators up to 16-18 Fr according to patient age
  Arms: childhood urolithiasis treated with mini PCNL Procedure
Procedure: RIRS procedure — RIRS Technique the 9.5 Fr ureteral access sheath (UAS). UAS was inserted over the guide wire under fluoroscopy control. A flexible ureteroscope was passed through the UAS. If the UAS did not pass over the guide wire, the investigator moved the flexible ureteroscopy over the guide wire without access sheat
  Arms: childhood urolithiasis treated with RIRS Procedure

SUMMARY:
The goal of this [ type of study:]prospective randomized clinical trial. The main question is to compare the outcomes of mini-percutaneous nephrolithotomy (m-PCNL) and retrograde intrarenal surgery (RIRS) in treating upper urinary tract calculus in children ≤ 10 years.

DETAILED DESCRIPTION:
With the increase in morbidity and incidence of pediatric kidney stone disease, childhood urolithiasis has become a significant health problem worldwide, especially in developing countries. Children with urinary calculi are at high risk for recurrent stone formation and may require multiple surgical interventions.

In recent decades, with the improvement of miniaturization of surgical equipment, the management of pediatric kidney stone disease has changed dramatically. As a result of these improvements, minimally invasive techniques, such as percutaneous nephrolithotomy (PCNL) and retrograde intrarenal surgery (RIRS) are alternative treatment options for children with upper urinary tract calculus.

Extracorporeal shock wave lithotripsy (ESWL) has been used for the treatment of upper urinary tract calculus < 2 cm. but, The significantly lower stone-free rates (SFR) of SWL as compared to the PCNL and RIRS, requirement for anesthesia, the possibility of parenchymal damage to the growing kidney and the need for additional sessions are the significant limitations of SWL

Mini-percutaneous nephrolithotomy (Mini-PCNL) is an adjustment of the standard PCNL procedure after the development of small-caliber instruments that has several advantages such as a smaller skin incision, smaller tract size, and less bleeding. However, mini-PCNL may cause severe complications because of fragile parenchyma, small caliber collecting system, and mobile kidney in pediatric patients.

with the persistent advancement of endoscopic instruments and flexible ureteroscope, the examination of the upper urinary tract has become more feasible, and retrograde intrarenal surgery (RIRS) can effectively compete with PCNL. However, the outcomes of the use of flexible ureteroscope in the pediatric population such as the risk of ureteral injury, stone-free rate especially in large stones (more than 2 cm), need for the ancillary procedure, the need to indwell double-J stent in advance and high cost of instrument and maintenance remain largely unknown, resulting in controversy about the clinical safety and efficacy of PCNL and RIRS in the treatment of upper urinary tract calculus.

In the current study, the investigators aimed to compare RIRS and mini-PCNL by evaluating The operative and postoperative outcomes for children ≤10 years of age with upper urinary tract calculus (1-2.5 cm).

ELIGIBILITY:
Inclusion Criteria:

* This study will include all children (age < 10 years) who undergo Mini-PCNL or RIRS with stone size (1_2.5 cm) for upper urinary tract stones

Exclusion Criteria:

* Children with urinary tract infections until treated
* Children with ureteral stricture
* Congenital urological anomalies
* Previous urological surgery

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
The fluoroscopy time of mini-PCNL and RIRS procedures in both groups | for each case in both groups the investigator assess the duration of fluoroscopy that the patient is exposed during the time of operation which range from (2-4 hours) through study completion, an average of 1.5 year"
  the duration of fluoroscopy time measured by seconds that the patient is exposed to during the procedure in both groups
the stone free rate in both groups | after one month from intervention
  Procedures will be accepted as stone free when there are no residual fragments or stone fragments <3 mm at follow-up CTUT
The operation time of mini-PCNL and RIRS procedures in both groups | for each case in both groups the investigator assess the time of operation from the induction of anesthesia till the end of operation "through study completion, an average of 1.5 year"
  the time of procedure measured by minutes in both groups
postoperative hospital stay time of mini-PCNL and RIRS procedures in both groups | or each case in both groups the investigator assess the hospital time from the day of admission of patient in hospital to do intervention till patient discharge from hospital through study completion, an average of 1.5 year"
  the post operative hospital stay measured by hours

CONTACTS AND LOCATIONS:
Overall Officials: mohamed sa salem, MD, Study Chair — Ain Shams University
Locations (1):
- Abdelrahman Nazmy Abbas Hatata, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu P, Song R, Yu Y, Yang J, Qi K, Tao R, Chen K, Zhang W, Gu M. Clinical efficacy of percutaneous nephrolithotomy versus retrograde intrarenal surgery for pediatric kidney urolithiasis: A PRISMA-compliant article. Medicine (Baltimore). 2017 Oct;96(43):e8346. doi: 10.1097/MD.0000000000008346. PMID 29069011
- [Background] Bastug F, Gunduz Z, Tulpar S, Poyrazoglu H, Dusunsel R. Urolithiasis in infants: evaluation of risk factors. World J Urol. 2013 Oct;31(5):1117-22. doi: 10.1007/s00345-012-0828-y. Epub 2012 Jan 19. PMID 22258667
- [Background] Gao X, Fang Z, Lu C, Shen R, Dong H, Sun Y. Management of staghorn stones in special situations. Asian J Urol. 2020 Apr;7(2):130-138. doi: 10.1016/j.ajur.2019.12.014. Epub 2019 Dec 30. PMID 32257806